CLINICAL TRIAL: NCT00003650
Title: Phase III Study of Combination Chemotherapy in Children With T Cell and Pre-B Cell Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy in Treating Children With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066742; FNCLCC-SFOP-96006-LMT-96; EU-98049
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Lymphoma
Keywords: stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Etoposide; Mercaptopurine; Methotrexate; Methylprednisolone; Mitoxantrone; Prednisone; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: etoposide
Drug: mercaptopurine
Drug: methotrexate
Drug: methylprednisolone
Drug: mitoxantrone hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase III trial to study the effectiveness of combination chemotherapy in treating children who have non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the event free survival at 2 and 5 years of children with T cell or pre-B cell non-Hodgkin's lymphoma treated with a sequential induction regimen, a consolidation regimen, a reintensification regimen, and a maintenance regimen.
* Assess the rate of local relapse at 2 and 5 years of these children after receiving this treatment.
* Determine the toxicity of this treatment in these patients.
* Determine the overall survival of these children at 5 years after receiving this treatment.

OUTLINE: This is a multicenter study.

Patients receive 5 weeks of induction chemotherapy consisting of prednisone IV twice a day on days 1-28, then decreasing in dose on days 29-35; vincristine IV on days 8, 15, 22, and 29; cyclophosphamide IV over 1 hour on day 8; daunorubicin IV over 24 hours on days 15, 22, and 29; asparaginase IV or IM on days 16, 18, 20, 23, 25, 27, 30, and 32; and methotrexate IV over 3 hours on day 8. Patients also receive methotrexate and methylprednisolone intrathecally (IT) on days 1, 4, 9, and 15.

Patients with a response over 50% proceed to 4-8 weeks of consolidation therapy. This regimen consists of vincristine IV on day 15, cyclophosphamide IV over 1 hour followed by methotrexate over 3 hours on day 1, cytarabine IV on days 2-5 and 8-11, asparaginase IV or IM on days 16 and 23, and methotrexate IV over 3 hours on day 15. Patients also receive methotrexate and methylprednisolone IT on days 2 and 16. Patients who achieve complete remission after 4 weeks repeat consolidation therapy for another course.

Patients then receive 4 weeks of interphase therapy consisting of oral mercaptopurine on days 1 and 22, methotrexate IV over 3 hours on days 1 and 15, and methotrexate and methylprednisolone IT on days 2 and 16.

Patients with pre-B cell lymphoma then proceed to maintenance therapy. Patients with T cell lymphoma proceed to reinduction therapy. Reinduction A is a 4 week course of chemotherapy administered during months 1, 3, and 5 and consists of vincristine IV on day 1; methotrexate IV over 3 hours on days 1, 8, 15, and 22; methotrexate and methylprednisolone IT on day 2; asparaginase IM or IV on day 2; and oral mercaptopurine. Reinduction B is also a 4 week course of therapy administered during months 2, 4, and 6. This consists of oral prednisone twice a day on days 1-5; cytarabine subcutaneously twice a day on days 1-4; methotrexate IV on days 1, 8, 15, and 22; and oral mercaptopurine.

Patients then proceed to maintenance therapy, which consists of methotrexate and mercaptopurine once a week. Patients with stage I, II, or III disease continue maintenance therapy for 18 months, while patients with stage IV disease continue this therapy for 24 months.

Patients with stage IV disease with neuromeningeal involvement receive triple intrathecal therapy consisting of methotrexate, cytarabine, and methylprednisolone, then reinduction A for months 1, 2, and 3, then reinduction B for months 4, 5, and 6 (if T cell lymphoma). These patients also receive cerebral irradiation during months 4 and 5. Patients with pre-B cell disease receive cerebral irradiation after intensification therapy.

Patients with less than 50% response after induction therapy or incomplete remission after 4-8 weeks of consolidation therapy, or who have a recurrence of disease are treated with the "VANDA" regimen consisting of dexamethasone on days 1-5; cytarabine over 3 hours twice a day on days 1 and 2; mitoxantrone IV over 1 hour on days 3 and 4; etoposide IV over 1 hour on days 3-5; and asparaginase IV over 1 hour or IM on days 7, 9, 11, and 13. Patients also receive triple intrathecal therapy (methotrexate, cytarabine, and methylprednisolone) on day 5.

Patients are followed every 2 months for 1 year, every 3 months for 2 years, every 4 months for 1 year, every 6 months for 1 year, then annually thereafter.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and/or cytologically confirmed T cell or pre-B cell non-Hodgkin's lymphoma

  * Lymphoblastic or peripheral T cell
  * Stage I, II, III, or IV
* No anaplastic lymphoma, large cell lymphoma, or small noncleaved cell lymphoma

PATIENT CHARACTERISTICS:

Age:

* 18 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No prior malignancy
* No chronic medical or psychological condition
* No congenital immunodeficiency
* HIV and HTLV negative
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior corticosteroids allowed

Radiotherapy:

* Not specified

Surgery:

* No prior organ transplant

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 179 (Actual)
Dates: Start 1997-02 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Bergeron, Study Chair — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France

REFERENCES:
- [Background] Ducassou S, Ferlay C, Bergeron C, Girard S, Laureys G, Pacquement H, Plantaz D, Lutz P, Vannier JP, Uyttebroeck A, Bertrand Y. Clinical presentation, evolution, and prognosis of precursor B-cell lymphoblastic lymphoma in trials LMT96, EORTC 58881, and EORTC 58951. Br J Haematol. 2011 Feb;152(4):441-51. doi: 10.1111/j.1365-2141.2010.08541.x. Epub 2011 Jan 7. PMID 21210776